CLINICAL TRIAL: NCT05528042
Title: Validation of the Performance of the COBOX Solution for Measuring Heart Rate and Respiratory Rate
Acronym: COBOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Quantiq.io (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A00818-35
Record Dates: First submitted 2022-08-31; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Anyone Who Meets the Eligibility Criteria Can Use the Software
Keywords: Heart rate, respiratory rate, COBOX
MeSH Terms: interventions — Heart Rate

STUDY DESIGN:
Intervention Model Description: We carry out a multicentric, prospective clinical research, evaluating the performance of the COBOX device to the extent and within the framework of usual care. Heart rate and respiratory rate are measured when a patient arrives in the emergency room, also, given the high attendance of these services, it seemed to us to be an excellent place for this study. This measurement is carried out as part of the patient's care pathway using the reference process techniques for taking measurements via a CE marked device and a manual counting reference method. The inclusions of the patient consultant in the emergencies service allow you to quickly obtain a large number of inclusions, and also, a great variability of the constants revealed by the different pathological stages. This allows a large reproduction in the combination of clinical situations and allows validating the actions in different contexts
Masking Description: All the parties will be aware of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N/A, only one arm (Other): All the patients that would like to participate and those where the inclusion criteria are past, are available to make the test. No drugs are administered.
  Interventions: Other: Heart rate and respiratory rate measurement

INTERVENTIONS:
Other: Heart rate and respiratory rate measurement — Validation of the performance of the heart rate (HR) measurement using COBOX medical device compared to a measurement carried out by applying the reference processes for taking measurements via a CE marked device.
  Evaluation of the performance of the respiratory rate (RR) measurement using COBOX medical device compared to a measurement carried out by a reference method of manual counting

SUMMARY:
Quantiq.io "COBOX" is a software as a medical device. It relies on remote photoplethysmography, allowing for the remote measurement of a patient's physiological parameters from a healthcare professional's or patient's device which can be a smartphone, a computer or a health station with an optical camera.

Quantiq.io software is a medical device which is :

contactless for the measurement non-invasive for the patient

In order to meet safety and quality standards, new health technologies require rigorous clinical validation with measurement performance at least equivalent to that of one CE marking measure device.

In this context, we assume that the COBOX device will take measurements of heart and respiratory rates equivalent to those taken by medical devices and current practices.

DETAILED DESCRIPTION:
The planned procedure is:

1. Oral information to the patient about the test by the nursing staff.
2. Patient signs the consent.
3. Collection of the patient's age, gender and Fitzpatrick phototype.
4. Collection of the patient identification number.
5. The nursing staff installs the oximeter on the patient's finger.
6. The nursing staff starts COBOX and begins to count the patient's breath in parallel
7. After 15, a first measurement is made by COBOX. The pulse oximeter reference result is acquired in parallel.
8. After 20s (5s after the previous measurement) a second measurement is made by COBOX.
9. After 25s (5 after the previous measurement) a third measurement is made by COBOX.
10. After 30s, the nursing staff enters the number of patient's breaths counted since the start.

The performance of the tool will be estimated by the concordance between the measurements obtained from the application of the reference technical process via a CE marked device and with the measurements obtained by COBOX.

An intraclass correlation coefficient (ICC) with its 95% confidence interval (95% CI) will be calculated. Measurement errors will be calculated and expressed as a percentage (root mean square error, etc.).

The two study samples will be compared by Student's t test and Fischer's F, with a desired significance for P value = 0.05, for all the analyses.

A DIXON test will be performed to assess the presence of statistically outliers within the samples.

These data will enable the COBOX tool, a class IIA medical device, to be validated in terms of measurement performance compared to a CE-marked device used in a reference technical process for taking measurements and a reference method for manual counting.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (older than 18 years old)
* Patient consulting in the emergency department of a participating center
* Patient having constant FC and FR taken by the reception organizing nurse (IOA) in the area dedicated to the reception of patients
* Patient who gave their consent to participate in the study

Exclusion Criteria:

* Patient in a state of vital emergency with direct entry into emergency service or intensive care
* Patient unable to express consent.
* Patient unable, for health reasons, to be face of COBOX.
* Patient unable to stay for 30 seconds facing the Cobox solution.
* Patient with skin stigma over more than 50% of the face (burn, graft)
* Patient with the face covered or not allowing access to the entire face (clothing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 323 (Estimated)
Dates: Start 2022-09-09 (Estimated); Primary Completion 2022-09-19 (Estimated); Study Completion 2022-09-19 (Estimated)

PRIMARY OUTCOMES:
Heart rate | less than 30 minutes
  validate the performance of the measurement of the heart rate (HR) measured by the COBOX medical device compared to a measurement carried out by applying the reference processes for taking measurements via a CE marked device.

SECONDARY OUTCOMES:
Respiratory rate | less than 30 minutes
  Evaluate the performance of the measurement of the respiratory rate (RR) measured by the COBOX medical device compared to a measurement carried out by a reference method of manual counting

IPD SHARING:
Plan to Share IPD: Yes
The information about the test is communicated by the nurse and if necessary completed by a doctor. This information must make it possible to answer all the patient's questions concerning the objective, the nature of the constraints, the foreseeable risks and the expected benefits of the research. It also specifies the patient's rights in the context of a clinical investigation and respects the eligibility criteria. A copy of the electronic consent form is then given to the patient by the investigating doctor.
Supporting Information: ICF
Time Frame: 09-19-2022
Access Criteria: Criteria:The consent form is electronic and must be signed before data can be provided for research. After electronic acceptance of the consent, a copy of the consent form is sent to the patient with his identification number allowing him at any time to ask the promoter to delete his data. For his part, the promoter only has access to the patient's identification number but his email address is not stored.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT05528042/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT05528042/ICF_001.pdf